CLINICAL TRIAL: NCT03037229
Title: Smartphone Twelve Lead Electrocardiogram Utility In ST-Elevation Myocardial Infarction
Acronym: ST LEUIS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: AliveCor (Industry)
Responsible Party: Principal Investigator, Gregory W. Barsness, Consultant, Assistant Professor of Medicine, Mayo Clinic
Other Study IDs: 16-004793
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: STEMI
Keywords: Myocardial Infarction; Ischemia; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Ischemia; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- STEMI: Subjects in which a STEMI protocol has been initiated.
  * An attempt will be made to do the standard 12-lead ECG first, followed immediately after by the Smartphone ECG
  * If the initial standard 12-lead ECG was already obtained, such as when the patient was first diagnosed with STEMI, a repeat ECG will be performed at the same time as the Smartphone ECG
  * If possible, the two ECGs will be taken in the Emergency Department, the critical care unit (CCU), or the catheterization laboratory just prior to cardiac catheterization. If not, then the two ECG's will be taken just after the cardiac catheterization is completed (i.e., within one hour of the procedure) while the patient is still in the catheterization laboratory and waiting for transport to the CCU
  * Both ECGs will be sent to the designated ECG reading station, to be read and evaluated by three independent cardiologists
  Interventions: Device: Smartphone ECG; Device: Standard 12-lead ECG
- Chest Pain: Subjects presenting at the emergency department with chest pain.
  * An attempt will be made to do the standard 12-lead ECG first, followed immediately after by the Smartphone ECG
  * If the initial standard 12-lead ECG was already obtained, such as when the patient was first diagnosed with STEMI, a repeat ECG will be performed at the same time as the Smartphone ECG
  * If possible, the two ECGs will be taken in the Emergency Department, the critical care unit (CCU), or the catheterization laboratory just prior to cardiac catheterization. If not, then the two ECG's will be taken just after the cardiac catheterization is completed (i.e., within one hour of the procedure) while the patient is still in the catheterization laboratory and waiting for transport to the CCU
  * Both ECGs will be sent to the designated ECG reading station, to be read and evaluated by three independent cardiologists
  Interventions: Device: Smartphone ECG; Device: Standard 12-lead ECG

INTERVENTIONS:
Device: Smartphone ECG
  Other Names: AliveCor Kardia Heart Monitor
Device: Standard 12-lead ECG

SUMMARY:
Is the Smartphone ECG (electrocardiogram) an acceptable replacement for a standard ECG in the identification of STEMI (ST Elevation Myocardial Infarction).

DETAILED DESCRIPTION:
The primary objective of this study is to determine if the Smartphone electrocardiogram (ECG) is an acceptable replacement for a standard ECG in the identification of ST Elevation Myocardial Infarction (STEMI).

Toward this objective, this study involves the following:

Obtain simultaneous recordings of a standard 12-lead ECG and the iPhone "12-lead equivalent" ECG on patients presenting with chest pain in which the STEMI protocol was activated.

Obtain simultaneous recordings of a standard 12-lead ECG and the iPhone "12-lead equivalent" ECG on patients presenting to the Emergency Department for evaluation of chest pain, not necessarily presenting with STEMI.

Reading of ECGs (standard 12-lead and iPhone) by three independent cardiologists, who are blinded to the initial clinical ECG readings, the type of ECG equipment used, and the patient's clinical information.

Assess the operational feasibility of using the Smartphone to obtain "12-lead equivalent" ECG recordings in patients suspected to have STEMI, and

Determine the possibility of pooling the data obtained from this study with data from other institutions conducting identical studies, and developing a future and statistical analysis plan to compare the sensitivity, specificity, positive predictive value and the negative predictive power of the iPhone ECG, using a paired standard 12-lead ECG as the gold standard.

There will be no therapeutic interventions. A single research-related procedure will be required, i.e., an iPhone ECG. Effort will be made to ensure that the performance of this procedure will not delay any treatment and/or diagnostic procedures that are part of usual or specialized care that the patient requires.

The individual patient's participation in the study will actually be only one day, i.e., the day the informed consent is obtained and the two comparison ECGs will be done.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures (patient or legally acceptable representative).
* Symptoms of chest pain upon presentation

Exclusion Criteria:

* Inability or refusal of the patient and/or the patient's legally-acceptable representative to provide written informed consent for any reason.
* Other conditions that in the opinion of the Principal Investigator or Co-Investigator(s) may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients, >18 years old, who are seen for chest pain, and/or patients for whom the STEMI protocol has been activated, will be screened for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Number of patients for whom the diagnoses (STEMI vs. non-STEMI) was in agreement between the standard 12-lead ECG and the iPhone "12-lead equivalent" ECG. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gregory W Barsness, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No